CLINICAL TRIAL: NCT02585167
Title: Endoscopic or Surgical Treatment of Complex Perianal Fistula. A Randomized Controlled Clinical Study
Brief Title: Endoscopic Treatment of Complex Anal Fistulas
Acronym: VAAFT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The significantly higher recurrence rate in the intervention group led to a serious ethical consideration of a premature closing of the study which was decided due to safety and benefit concerns
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Karam Matlub Sørensen, læge, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-20150053
Record Dates: First submitted 2015-10-20; First posted 2015-10-23 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Anal Fistula
Keywords: VAAFT; anal fistula; sphincter reconstruction
MeSH Terms: conditions — Rectal Fistula | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Operation (Active Comparator): the fistula will be excised after dividing the sphincter and primary reconstruction
  .
  Interventions: Procedure: operation
- VAAFT (Experimental): the fistula tract will be visualized by scope, closing the internal opening with absorbable sutures.
  Interventions: Device: VAAFT

INTERVENTIONS:
Procedure: operation — the fistula will be excised after dividing the sphincter and primary reconstruction will be performed with absorbable sutures, closing the internal opening and leaving the external opening unclosed for drainage.
  Other Names: Fistulectomy and primary sphincter reconstruction
  Arms: Operation
Device: VAAFT — Karl Storz Video Equipment is used. The fistula tract will be visualized from the external to the internal opening, closing the internal opening with absorbable sutures, then brushing and cauterization of the tract(s) leaving the external opening unclosed for drainage.
  Arms: VAAFT

SUMMARY:
This is a randomised controlled trial to evaluate the outcome of treatment of complex perianal fistula by Video-assisted anal fistula treatment (VAAFT) compared to fistulectomy and sphincter reconstruction as standard surgical procedure.

DETAILED DESCRIPTION:
The surgical treatment of complex fistulas is difficult and ideally aims to completely heal the fistula and prevent recurrence without affecting the anal sphincter function. The definitive surgical treatment options include transsphincteric fistulectomy and sphincter repair, intersphincteric ligation of the fistula tract (LIFT), transanal advancement flap and cutting Seton suture. All the methods caries a relative high recurrence and complication rate including the risk of anal incontinence .Transsphincteric fistulectomy and primary reconstruction of the anal sphincter has been reported to have a healing rate between 90 - 95,8 %, recurrence rate of 7,1-9,7 % and 5-30 % experience incontinence in varying degree. Video-assisted anal fistula treatment (VAAFT) is a novel sphincter saving procedure for treating complex anal fistulas and recently introduced with promising early results with a healing rate of 74-87.1 % after 1 year. The procedure can be done as a day-case surgery with the ability of precise identification of the fistula tract, including the presence of secondary branches. The method includes an endoscopic debridement and closure of the internal opening. Only few scientific reports of the method has been published and only with short term results, and there is a need of validating the efficacy of this procedure in a prospective randomized trial. There are few randomised controlled trials in the literature on the treatment of complex anal fistulas treatment and there is no conclusive evidence of which method is the best. Furthermore the knowledge of changes in quality of life and functional results in terms of standardized continence evaluation and manometric studies are either contradictive or simply lacking after the surgery for anal fistulas. The aim of this study is to conduct a randomized clinical trial to compare VAAFT (mini invasive and sphincter-saving) with the traditional transsphincteric fistulectomy and primary reconstruction in terms of recurrence rate, manometric and functional changes as well as changes in quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complex transsphincteric anal fistulas >18 yrs old.

Exclusion Criteria:

* Crohns fistulas
* Signs of suppuration or/and branching.
* Malignancy within 5 yrs.
* Previous radiotherapy of the abdomen and pelvis.
* Current Immune- suppressive treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
The recurrence rate of perianal fistula | 6 months
  A comparison on the rate of recurrence of anal fistula in each group will be performed by t-test. A p-value of less than 0.05 will be considered as statistical significant.

SECONDARY OUTCOMES:
changes in quality of life score | baseline and 6 months
  A comparison on changes in quality of life, using The Short Form (36) Health Survey in each group will be performed by t-test. A p-value of less than 0.05 will be considered as statistical significant.
changes in fecal incontinence score | baseline and 6 months
  A comparison on changes in Wexner score in each group will be performed by t-test. A p-value of less than 0.05 will be considered as statistical significant.
changes in manometric study | baseline and 6 months
  A comparison on changes in manometric study(including maximum resting pressure, maximum squeeze pressure) in each group will be performed by t-test. A p-value of less than 0.05 will be considered as statistical significant.

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Background] Barwood N, Clarke G, Levitt S, Levitt M. Fistula-in-ano: a prospective study of 107 patients. Aust N Z J Surg. 1997 Feb-Mar;67(2-3):98-102. doi: 10.1111/j.1445-2197.1997.tb01911.x. PMID 9068549
- [Background] Nicholls J. Anal fistula. Colorectal Dis. 2012 May;14(5):535. doi: 10.1111/j.1463-1318.2012.03025.x. No abstract available. PMID 22469475
- [Background] Lundby L, Hagen K, Christensen P, Buntzen S, Thorlacius-Ussing O, Andersen J, Krupa M, Qvist N. Treatment of non-IBD anal fistula. Dan Med J. 2015 May;62(5):C5088. PMID 26050835
- [Background] Steele SR, Kumar R, Feingold DL, Rafferty JL, Buie WD; Standards Practice Task Force of the American Society of Colon and Rectal Surgeons. Practice parameters for the management of perianal abscess and fistula-in-ano. Dis Colon Rectum. 2011 Dec;54(12):1465-74. doi: 10.1097/DCR.0b013e31823122b3. No abstract available. PMID 22067173
- [Background] Hvas CL, Dahlerup JF, Jacobsen BA, Ljungmann K, Qvist N, Staun M, Tottrup A. Diagnosis and treatment of fistulising Crohn's disease. Dan Med Bull. 2011 Oct;58(10):C4338. PMID 21975159
- [Background] Nicholls RJ. Fistula in ano: an overview. Acta Chir Iugosl. 2012;59(2):9-13. doi: 10.2298/aci1202009n. PMID 23373352
- [Background] Christiansen J, Moesgaard FA. [Treatment of anal fistulas]. Ugeskr Laeger. 2002 Sep 23;164(39):4519-21. No abstract available. Danish. PMID 12380393
- [Background] Bokhari S, Lindsey I. Incontinence following sphincter division for treatment of anal fistula. Colorectal Dis. 2010 Jul;12(7 Online):e135-9. doi: 10.1111/j.1463-1318.2009.01872.x. Epub 2009 Apr 10. PMID 19486093
- [Background] Ratto C, Litta F, Parello A, Zaccone G, Donisi L, De Simone V. Fistulotomy with end-to-end primary sphincteroplasty for anal fistula: results from a prospective study. Dis Colon Rectum. 2013 Feb;56(2):226-33. doi: 10.1097/DCR.0b013e31827aab72. PMID 23303152
- [Background] Roig JV, Garcia-Armengol J, Jordan JC, Moro D, Garcia-Granero E, Alos R. Fistulectomy and sphincteric reconstruction for complex cryptoglandular fistulas. Colorectal Dis. 2010 Jul;12(7 Online):e145-52. doi: 10.1111/j.1463-1318.2009.02002.x. Epub 2009 Jul 9. PMID 19604292
- [Background] Perez F, Arroyo A, Serrano P, Sanchez A, Candela F, Perez MT, Calpena R. Randomized clinical and manometric study of advancement flap versus fistulotomy with sphincter reconstruction in the management of complex fistula-in-ano. Am J Surg. 2006 Jul;192(1):34-40. doi: 10.1016/j.amjsurg.2006.01.028. PMID 16769272
- [Background] Roig, Garcia-Armengol, Jordan, Alos, Solana. Immediate reconstruction of the anal sphincter after fistulectomy in the management of complex anal fistulas. Colorectal Dis. 1999 May;1(3):137-40. doi: 10.1046/j.1463-1318.1999.00021.x. PMID 23577759
- [Background] Jivapaisarnpong P. Core out fistulectomy, anal sphincter reconstruction and primary repair of internal opening in the treatment of complex anal fistula. J Med Assoc Thai. 2009 May;92(5):638-42. PMID 19459524
- [Background] Tobisch A, Stelzner S, Hellmich G, Jackisch T, Witzigmann H. Total fistulectomy with simple closure of the internal opening in the management of complex cryptoglandular fistulas: long-term results and functional outcome. Dis Colon Rectum. 2012 Jul;55(7):750-5. doi: 10.1097/DCR.0b013e3182569b29. PMID 22706126
- [Background] Meinero P, Mori L. Video-assisted anal fistula treatment (VAAFT): a novel sphincter-saving procedure for treating complex anal fistulas. Tech Coloproctol. 2011 Dec;15(4):417-22. doi: 10.1007/s10151-011-0769-2. Epub 2011 Oct 15. PMID 22002535
- [Background] Meinero P, Mori L, Gasloli G. Video-assisted anal fistula treatment: a new concept of treating anal fistulas. Dis Colon Rectum. 2014 Mar;57(3):354-9. doi: 10.1097/DCR.0000000000000082. PMID 24509459
- [Background] Schwandner O. Video-assisted anal fistula treatment (VAAFT) combined with advancement flap repair in Crohn's disease. Tech Coloproctol. 2013 Apr;17(2):221-5. doi: 10.1007/s10151-012-0921-7. Epub 2012 Nov 23. PMID 23179892
- [Background] Zbar AP. "Video-assisted anal fistula treatment (VAAFT): a novel sphincter-saving procedure to repair complex anal fistulas" by Piercarlo Meinero and Lorenzo Mori. Tech Coloproctol. 2011 Dec;15(4):423-4. doi: 10.1007/s10151-011-0771-8. No abstract available. PMID 22016156
- [Background] Quah HM, Tang CL, Eu KW, Chan SY, Samuel M. Meta-analysis of randomized clinical trials comparing drainage alone vs primary sphincter-cutting procedures for anorectal abscess-fistula. Int J Colorectal Dis. 2006 Sep;21(6):602-9. doi: 10.1007/s00384-005-0060-y. Epub 2005 Nov 30. PMID 16317550
- [Background] Grucela A, Gurland B, Kiran RP. Functional outcomes and quality of life after anorectal surgery. Am Surg. 2012 Sep;78(9):952-6. PMID 22964203
- [Background] Kasparek MS, Glatzle J, Temeltcheva T, Mueller MH, Koenigsrainer A, Kreis ME. Long-term quality of life in patients with Crohn's disease and perianal fistulas: influence of fecal diversion. Dis Colon Rectum. 2007 Dec;50(12):2067-74. doi: 10.1007/s10350-007-9006-5. PMID 17680311
- [Background] Riss S, Schwameis K, Mittlbock M, Pones M, Vogelsang H, Reinisch W, Riedl M, Stift A. Sexual function and quality of life after surgical treatment for anal fistulas in Crohn's disease. Tech Coloproctol. 2013 Feb;17(1):89-94. doi: 10.1007/s10151-012-0890-x. Epub 2012 Sep 6. PMID 22956209
- [Background] Roig JV, Jordan J, Garcia-Armengol J, Esclapez P, Solana A. Changes in anorectal morphologic and functional parameters after fistula-in-ano surgery. Dis Colon Rectum. 2009 Aug;52(8):1462-9. doi: 10.1007/DCR.0b013e3181a80e24. PMID 19617761
- [Background] Ha HT, Fleshman JW, Smith M, Read TE, Kodner IJ, Birnbaum EH. Manometric squeeze pressure difference parallels functional outcome after overlapping sphincter reconstruction. Dis Colon Rectum. 2001 May;44(5):655-60. doi: 10.1007/BF02234561. PMID 11357023
- [Background] Sailer M, Bussen D, Debus ES, Fuchs KH, Thiede A. Quality of life in patients with benign anorectal disorders. Br J Surg. 1998 Dec;85(12):1716-9. doi: 10.1046/j.1365-2168.1998.00958.x. PMID 9876082
- [Background] Parks AG, Gordon PH, Hardcastle JD. A classification of fistula-in-ano. Br J Surg. 1976 Jan;63(1):1-12. doi: 10.1002/bjs.1800630102. PMID 1267867
- [Derived] Sorensen KM, Moller S, Qvist N. Video-assisted anal fistula treatment versus fistulectomy and sphincter repair in the treatment of high cryptoglandular anal fistula: a randomized clinical study. BJS Open. 2021 Sep 6;5(5):zrab097. doi: 10.1093/bjsopen/zrab097. PMID 34611700
- See also: OPEN homepage — http://open.rsyd.dk/OpenProjects/da/openProject.jsp?openNo=145